CLINICAL TRIAL: NCT07376096
Title: Diagnostic and Prognostic Value of Liquid Biopsy in Germ Cell Tumors
Brief Title: Liquid Biopsy in Germ Cell Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: FWF - Österreichischer Wissenschaftsfonds (Unknown); Medical University of Innsbruck (Unknown); Medical University of Vienna (Other); Klinikum Ottakring Vienna (Unknown); Klinikum Favoriten Vienna (Unknown); Klinikum Klagenfurt am Wörthersee (Other); Landeskrankenhaus Salzburg (Unknown); Johannes Kepler Universität Linz (Unknown); Cantonal Hospital of St. Gallen (Other); Kantonsspital Graubünden (Other); Luzerner Kantonsspital (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Düsseldorf (Other); Vivantes Klinikum Am Urban, Berlin (Unknown); Universitätsklinikum Krems (Unknown); Universitätsklinikum Wiener Neustadt (Unknown)
Responsible Party: Sponsor
Other Study IDs: KLP9070624_4
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: 100 Stage I Patients; 100 Metastatic Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA and microRNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage I: non-metastatic testicular germ cell tumors
- Stage II-III: metastatic testicular germ cell tumors

SUMMARY:
Theoretical framework: Testicular germ cell tumors (TGCT) are characterized by frequent chromosomal anomalies such as gain of chromosome 12p and low rates of somatic mutations. Cell-free circulating tumor DNA (ctDNA) has been investigated in some cancers but only a few studies explored the presence of ctDNA in TGCT. The consistent gain of genetic material from chromosome 12p makes TGCT patients to ideal candidates for liquid biopsy investigations. We have analyzed three pre-chemo samples with our plasma-Seq approach and applied the ichorCNA algorithm to call for somatic copy number alterations (SCNA) and estimate the tumor fraction. Besides the frequently observed chromosome 12p gain, a variety of other SCNA were detected indicating that shallow whole genome sequencing (sWGS) is a suitable approach to analyze ctDNA in TGCT. Only 60% of TGCT patients express the classical markers alpha fetoprotein (AFP) and beta (human chorionic gonadotropin) HCG. Biomarkers to monitor patients who don't express the classical markers are of great need.

Hypotheses: We postulate that tumor-specific aberrations can be detected non-invasively in plasma DNA from patients with metastatic TGCT and serve as a diagnostic tool. Furthermore, we will investigate if the change of ctDNA during curative treatment can be used as monitoring tool and allows risk classification in comparison to conventional markers and the novel micro RNA biomarker miR-371a-3p (prognostic value of ctDNA).

Methods: For ctDNA and micro RNA analysis, blood samples will be drawn from patients before orchiectomy, before chemotherapy start, prior to the second cycle of chemotherapy, after completion of treatment and in case of relapse. In order to identify SCNA and to estimate the tumor content in plasma we will employ sWGS and analyze the data with the ichorCNA algorithm for a detection of SCNA. Since TGCT have low rates of somatic mutations, orchiectomy samples from patients with disease recurrence and plasma samples at time of recurrence will also be compared with the Biomodal platform which allows analysis of genetic as well as epigenetic changes.

DETAILED DESCRIPTION:
Study design This is a prospective, non-therapeutic trial to test the diagnostic and prognostic value of ctDNA in TGCT patients. 100 patients with metastatic TGCT presenting to treating centers in Austria, centers from the SAG registry and selected centers from Germany will be asked to participate and blood will be drawn for ctDNA and miR-371a-3p analysis during the course of disease at defined time points. In addition, 100 patients with stage I disease within Austria will be included.

Sampling Prior to surgery and intraoperative: Plasma and micro RNA samples will also be obtained prior to surgery. Plasma will be also obtained intraoperatively form the testicular vein.

After orchiectomy (before the 1st cycle of chemotherapy): Blood will be drawn into two PAXgene® Blood ccfDNA tubes (approx. 20ml) for ctDNA analysis before the start of chemotherapy. PAXgene tubes and tumor tissue will be send and stored at the Biobank of the Medical University of Graz. For the miR-371a-3p collection 10ml blood will be collected in serum tubes, centrifuged and 2ml serum stored at -80°.

Before the second cycle of chemotherapy: To evaluate treatment response with ctDNA levels, two PAXgene® Blood ccfDNA tubes (approx. 20ml) will be collected before the application of the second chemotherapy cycle. For the miR-371a-3p collection 10ml blood will be collected and processed as described above.

After completion of treatment: When the patient has completed first line treatment another two PAXgene® Blood ccfDNA tubes (approx. 20ml) will be drawn for ctDNA analysis. For the miR-371a-3p collection 10ml blood will be collected and processed as described above.

At the time of relapse: Approximately 20-30% of patients with metastatic TGCT will relapse. These can be primarily non-responders or patients who relapse after completion of chemotherapy which usually occurs within two years. Two PAXgene® Blood ccfDNA tubes (approx. 20ml) will be drawn for ctDNA analysis at the time of relapse (evident on imaging or rise of classical tumor markers). For the miR-371a-3p collection 10ml blood will be collected.

Sample analysis Comprehensive molecular profiling of the primary tumor tissue DNA from tumors samples will be isolated using the GeneRead DNA FFPE Kit (QIAGEN). DNA will be quantified using the Qubit (Thermo Fisher). To comprehensively profile tissues the duet multiomics solution evoC platform will be used, which not only interrogates the genome with respect to genetic alterations, but also enables epigenetic analysis differentiating between methylcytosine (mC) and hydroxymethylcytosine (hmC). Such a combined genome and methylome may reveals a correlation in 5mC and 5hmC by distinguishing between the two within regions of open chromatin and gene expression. The same data set can be used to infer genome-wide copy alterations. SCNA and focal alterations will be called using established in-house algorithms. Tumor purity/ploidy will be assessed using the ichorCNA algorithm, a hidden Markov model (HMM) for the probabilistic modeling and works in sequencing coverages down to 0.1X and enables a detection of SCNA down to a tumor fraction of 3%. In case the clonality of the tumor tissue is too low, exomes sequencing will be optionally performed for deep mutation profiling. Biomodal data from tissues will be compared to plasma samples from the time point of progression as well as to chemosensitive tumors to identify factors contributing to acquired and primary resistance. Tissue collected during surgery will be send to the department of pathology at the Medical University of Graz where DNA isolation and genome sequencing will be performed.

Analysis of ctDNA Blood will be collected in PAXgene® Blood ccfDNA and sent to the Institute of Human Genetics for further processing. cfDNA extraction from plasma will be performed using the QIAsymphony PAXgene Blood ccfDNA Kit (QIAGEN). To identify SCNA, we will employ sWGS (plasma-Seq) and again analyze the data with the ichorCNA algorithm. Alternatively, dPCR will be performed to screen for the 12p gain to increase the sensitivity. Plasma samples with a high tumor fractions from patients with disease recurrence will be additionally analyzed using the Biomodal platform and whole exome sequencing. Genetic and epigenetic profiles will be compared to the diagnostic tissue gained from orchiectomy. We have already successfully implemented the Biomodal platform in our lab in the framework of prostate cancer project. Moreover, we have evaluated an ctDNA-specific exome enrichment kit, which enables reliable variant detection down to 1%. All bioinformatics tools to analyze exome and Biomodal data sets are well established at the Institute of Human Genetics of the Medical University of Graz.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with the age ≥ 18years with
* Seminomatous or non-seminomatous germ cell tumors (extragonadal origin is allowed)
* Metastatic disease
* Stage I patients on active surveillance (for seminoma patients at least one risk factor, rete testis infiltration or tumor size > 4cm, should be present)

Exclusion Criteria:

* Other tumors than germ cell tumors of the testis
* Patients with a second malignancy within the last 5 years (except germ cell tumors)
* Stage I patients who received adjuvant treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: We aim to recruit 200 testicular germ cell tumor patients, 100 subjects with metastatic disease and 100 patients with stage I disease.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-02-15 (Estimated); Study Completion 2030-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with detectable ctDNA | 2 years

SECONDARY OUTCOMES:
To compare the sensitivity and specificity of ctDNA with miR-371a-3p | 2 years

IPD SHARING:
Plan to Share IPD: Yes
The publication underlying data will be published in zenodo under a CC BY license.
  The data will get a DOI through data publication in zenodo and will be referenced in the publication´ s data availability statement.
Supporting Information: CSR